CLINICAL TRIAL: NCT00905086
Title: Psychosocial Adjustment During the Post-Radiation Treatment Transition
Brief Title: Psychosocial Adjustment After Radiation Therapy in Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE3Z08; P30CA043703 (NIH); CASE3Z08 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer; Cognitive/Functional Effects; Colorectal Cancer; Lung Cancer; Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: cognitive/functional effects; psychosocial effects of cancer and its treatment; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire administration — Two weeks before completing planned radiotherapy, patients undergo assessment of stress appraisal and other factors predictive of post-radiotherapy psychosocial adjustment. At 1 month after completion of radiotherapy, patients undergo repeat assessment of stress appraisal and psychosocial adjustment.
Procedure: cognitive assessment — Patients complete psychosocial assessments, including measures of patient perceptions of their illness (i.e., cognitive appraisal) and of the factors influencing their perceptions (i.e., uncertainty by the Mishel Uncertainty in Illness Scale-Community Form; symptom distress by the Memorial Symptom Assessment Scale Short Form; and comorbidity by the Charlson Comorbidity Index).
Procedure: psychosocial assessment and care — Patients complete psychosocial assessments, including measures of patient perceptions of their illness (i.e., cognitive appraisal) and of the factors influencing their perceptions (i.e., uncertainty by the Mishel Uncertainty in Illness Scale-Community Form; symptom distress by the Memorial Symptom Assessment Scale Short Form; and comorbidity by the Charlson Comorbidity Index).
Procedure: quality-of-life assessment — At 1 month after completion of radiotherapy, patients undergo repeat assessment of stress appraisal and psychosocial adjustment.

SUMMARY:
RATIONALE: Gathering information about psychological and social adjustment after radiation therapy in patients with cancer may help doctors plan the best treatment.

PURPOSE: This clinical trial is studying psychosocial adjustment after radiation therapy in patients with breast cancer, colorectal cancer, lung cancer, or prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To describe psychosocial adjustment after radiotherapy in patients with stage I, II, or III breast, colorectal, lung, or prostate cancer.
* To determine if cognitive appraisal of health predicts psychosocial adjustment of these patients after radiotherapy.
* To examine whether social support moderates the relationship between cognitive appraisal of health and psychosocial adjustment of these patients after radiotherapy.
* To examine whether self-efficacy for coping with cancer moderates the relationship between cognitive appraisal of health and psychosocial adjustment of these patients after radiotherapy.
* To measure the effect of symptom distress, uncertainty, medical factors, and personal factors on cognitive appraisal of health of these patients before ending radiotherapy.

OUTLINE: Two weeks before completing planned radiotherapy, patients undergo assessment of stress appraisal and other factors predictive of post-radiotherapy psychosocial adjustment. Patients complete psychosocial assessments, including measures of patient perceptions of their illness (i.e., cognitive appraisal) and of the factors influencing their perceptions (i.e., uncertainty by the Mishel Uncertainty in Illness Scale-Community Form; symptom distress by the Memorial Symptom Assessment Scale Short Form; and comorbidity by the Charlson Comorbidity Index). Measures of patient social support and self-efficacy for coping are also assessed. At 1 month after completion of radiotherapy, patients undergo repeat assessment of stress appraisal and psychosocial adjustment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast, colorectal, lung, or prostate cancer

  * Stage I, II, or III disease
  * Nonmetastatic disease
* Undergoing first course of curative radiotherapy, as indicated in the medical record

  * Receiving treatment as an outpatient
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Able to receive treatment as an outpatient
* Lives in northeastern Ohio
* Cognitively intact, as evidenced by orientation to person, place, and time
* Has a telephone
* No hearing impairment (must be able to hear instructions)
* No malignancy expected to require surgery or chemotherapy ≤ 2 months after treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy for another type of cancer
* No concurrent or planned chemotherapy or surgery for at least 2 months after radiotherapy
* No concurrent treatment for recurrent cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Relationship between stress appraisal (as assessed by CAHS at baseline) and psychosocial adjustment (as assessed by PAIS-SR at 1 month after radiotherapy) | one month after radiotherapy
Relationship between stress appraisal and uncertainty, symptom distress, cancer stage, comorbidities, age, gender, race/ethnicity, and education at 2 weeks prior to completing radiotherapy | 2 weeks prior to radiotherapy
Social support (as assessed by MOS-SSS) and self-efficacy (as assessed by CBI-L v2.0) as moderators of the relationship between cognitive appraisal and adjustment | At 1 month after completion of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Daly, PhD, RN, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center; Susan Mazanec, RN, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States